CLINICAL TRIAL: NCT05894382
Title: A Randomized Controlled Study on the Effectiveness, Safety and Adaptability of Double Helix Design Defocus Lens Spectacle Frames for Correction of Visual Acuity in Children and Adolescents, and Control of Myopia.
Brief Title: Double Helix Design Defocus Lens Spectacle (RACE) for Myopia Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230421v1.3
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-05

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Double Helix Design Defocus Lens Spectacle (RACE) for 2 years
  Interventions: Device: Double Helix Design Defocus Lens Spectacle (RACE)
- Group B (Placebo Comparator): 1. st year: single-vision spectacle lenses
  2. nd year: double helix design defocus lens spectacle (RACE)
  Interventions: Device: Double Helix Design Defocus Lens Spectacle (RACE); Device: single-vision spetacle lens

INTERVENTIONS:
Device: Double Helix Design Defocus Lens Spectacle (RACE) — Double Helix Design Defocus Lens Spectacle wearing more than 10h/day.
Device: single-vision spetacle lens — single-vision spetacle lens wearing more than 10h/day.
  Arms: Group B

SUMMARY:
This study uses 1.585 double helix defocus lens PC lenses with a unique optical design that includes a globally coherent visible area and complementary left and right helices that can form clear images. In addition, the helical arrangement and reduced slit area can generate defocusing signals, inhibiting the development of myopia. Therefore, based on previous research, this study plans to evaluate the safety and effectiveness of 1.585 double helix defocus lens PC frame eyeglasses in controlling the progression of myopia in children and adolescents through a randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Race: Chinese children and adolescents.
2. Age 6-13 years, gender unrestricted.
3. Cycloplegic refraction SER: -0.75DS~-5.0DS in both eyes.
4. Best corrected visual acuity of both eyes reaches 1.0 (0.00 logMAR 6/6).
5. Refractive astigmatism and astigmatism are no more than 1.5D.
6. During the study period, willing to wear glasses provided by the researcher only (>10 hours) and without additional interventions.
7. Willing to be randomly assigned.
8. Able to sign an informed consent form with the accompaniment and understanding of parents or guardians.

Exclusion Criteria:

1. Allergic or intolerant to medications used for ciliary muscle paralysis.
2. Received any nearsightedness treatment such as atropine, rigid gas permeable contact lens, bifocal/progressive lens, red light therapy, or acupuncture within 30 days before the study.
3. Received defocus lenses for nearsightedness treatment in the past.
4. Diagnosed with any eye disease other than nearsightedness, including strabismus (esotropia greater than 8 prism diopters or exotropia greater than 12 prism diopters), corneal diseases, conjunctival or eyelid damage or other conditions (such as keratoconus, herpes simplex keratitis, etc.).
5. History of eye surgery (including strabismus correction surgery).
6. Eye or systemic diseases that might be associated with nearsightedness or its progression, such as Marfan syndrome, retinopathy of prematurity, diabetes, etc.
7. Anatomical or dermatological factors that may interfere with the wearing of spectacle frames.
8. Other reasons that the researcher deems inappropriate for the participant to be included in the study, such as excessively high expectations for the effectiveness of defocus lenses, or plans to use other nearsightedness intervention strategies simultaneously with the study.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Estimated)
Dates: Start 2023-06-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Spherical Equivalent change | 1 year
  cycloplegic SE change

SECONDARY OUTCOMES:
Axial Length change | 1 year
Visual Acuity change | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangui He, Shanghai, Shanghai Municipality, China